CLINICAL TRIAL: NCT05855564
Title: Implementing a School-based Mindfulness Program in Primary School Curriculum
Brief Title: Implementing a School-based Mindfulness Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: School
Record Dates: First submitted 2023-04-03; First posted 2023-05-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-03

CONDITIONS: Mental Health Wellness 1
Keywords: student mental health; school-based mindfulness training; students with special needs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- School-based Mindfulness program (Experimental): Eight session of mindfulness-based program based on Mindfulness Matters developed by Eline Snel
  Interventions: Behavioral: mindfulness matters

INTERVENTIONS:
Behavioral: mindfulness matters — Classroom program will be provided to primary one students in eight primary schools and they will receive an 8 session mindfulness matters program, developed by Eline Snel, delivered by their teachers. Each session lasts for 30 minutes. The program includes mindfulness exercises, psychoeducation, discussion and sharing activities. For students with special needs, same programs will be delivered by teachers or social workers in small groups and each groups has 4 to 7 students. Program content is consistent with the classroom program.

SUMMARY:
The outcomes and implementation processes of the school based mindfulness program, as a universal prevention program in classroom as and support group programs for students with special education needs will be investigated. The study of classroom program will apply quasi-experimental design, comparing the pretest and posttest of seven primary schools with implementation of mindfulness programs with three schools with ordinary school activities only. A total of 800 students will be recruited to receive an eight session mindfulness program in classroom as a universal prevention program. Ten support group for students with special education needs will apply mindfulness programs, and its outcome will be evaluated using repeated time measures.

ELIGIBILITY:
Inclusion Criteria:

* students in participating schools
* students with parent's consent

Exclusion Criteria:

* student without parent's consent

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
positive self-perception | immediately before the intervention, and immediately after the intervention
  measured by Self-Evaluation Scale for Children. Values from 0 to 80. The higher the score, the stronger the positive self-perception

SECONDARY OUTCOMES:
peer relationship | before the intervention, and immediately after the intervention
  measured by Assessment Programme for Affective and Social Outcomes (2nd Version). Values from 6 to 24. The higher the score, the better the peer relationship
attitude towards school | before the intervention, and immediately after the intervention
  measured by Assessment Programme for Affective and Social Outcomes (2nd Version). Values from 6 to 24. The higher the score, the stronger the positive attitude towards school.
organized, nondisruptive, and nonimpulsive behaviors | before the intervention, and immediately after the intervention
  measured by Self-Evaluation Scale for Children. Values from 0 to 70. The higher the score, the higher the severity of problem behaviors
executive functioning | before the intervention, and immediately after the intervention
  measured by ratings of parent and teacher of Behavior Rating Inventory of Executive Function, second edition. The scale includes subscales in inhibit, self-monitor, behavior regulation, emotion regulation, cognitive regulation. The higher the score, the stronger the functioning.
creativity | before the intervention, and immediately after the intervention.
  measured by the Test for Creative Thinking-Drawing Production. The completed drawings are scored according to the following 10 criteria : (1) continuations, (2) completion, (3) new element, (4 ) connections made with a (5) connections made to produce a theme, (6) boundary breaking that is fragment dependent, (7) boundary breaking that is fragment independent, (8) perspective, (9) humour and affective, (10) unconventionality. The scores for all the criteria except unconventionality range d from 0 to 6. Each unconventionality criterion was score d either 0 or 3. The maximum score is 60. The higher the score, the higher the creativity.
self-regulation | before the intervention, and immediately after the intervention
  measured by The Head-Toes-Knees-Shoulders (HTKS) task
cortisol | before the intervention, and immediately after the intervention
  measured by salivary cortisol (this measure is administered for students with special needs only)

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong
  - Hong Kong Polytechnic University, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The funder decided not to share the data.